CLINICAL TRIAL: NCT05383313
Title: Psilocybin Versus Ketamine - Fast Acting Antidepressant Strategies in Treatment-resistant Depression
Brief Title: Psilocybin Versus Ketamine in Treatment-Resistant Depression
Acronym: PSIKET_001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Collaborators: Czech Health Research Council (Unknown); Czech Clinical Research Infrastructure Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: PSIKET_001CZE
Record Dates: First submitted 2021-09-07; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2021-09

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Psilocybin (Experimental): 25 mg, orally (capsule), single administration
  Interventions: Drug: Psilocybin
- Ketamine (Active Comparator): 250 mg, orally (capsule), single administration
  Interventions: Drug: Ketamine Hydrochloride
- Midazolam (Placebo Comparator): 5 mg, orally (capsule), single administration
  Interventions: Drug: Midazolam Ph. Eur 9.0

INTERVENTIONS:
Drug: Psilocybin — Effect of psilocybin on treatment-resistant depression
  Arms: Psilocybin
Drug: Ketamine Hydrochloride — Effect of ketamine on treatment-resistant depression
  Arms: Ketamine
Drug: Midazolam Ph. Eur 9.0 — Effect of midazolam on treatment-resistant depression
  Arms: Midazolam

SUMMARY:
The main goal is to compare the antidepressant effects of psilocybin and ketamine in patients with TRD versus the antidepressant inactive substance midazolam. The primary endpoint will be the antidepressant effect on the Montgomery- Asberg Depression Rating Scale (MADRS) 24 hours after treatment, the key secondary endpoints being the duration of antidepressant effect, the number of responses and remissions, and the time to standard antidepressant treatment during 3 months of observation. The exploratory part of the study aims to monitor changes in the functional brain states using simultaneous EEG / fMRI, before treatment versus 1 day and 1 week after. Based on literature data and recent data from healthy volunteers who participated in a previous study with psilocybin, the investigator will correlate antidepressant effects of drugs (using psychometric scales and reactions to emotionally salient stimuli (eye tracker)) with entropy and functional connectivity measures. Finally the investigator will explore the role of plasmatic neurobiological biomarkers in depression (BDNF, prolactin, ACTH and oxytocin).

DETAILED DESCRIPTION:
The main aim of the study is to verify the efficacy and safety of a single dose of psilocybin 20 mg in the treatment of TRD in adults in a randomized clinical trial with active comparator ketamine 200 mg (rapid onset acting antidepressant) and negative control midazolam 5 mg (drug with no antidepressant properties). Primary objective: 1) verification of the rapid antidepressant effect of psilocybin compared to ketamine using the MADRS scale at 24 hours. Secondary objectives: 1) on days 3, 7 and 14 and 3, 4, 5, 6, 8 and 12 weeks after application of the substances, evaluate / compare: a) the duration of effects of both substances using the MADRS scale b) antidepressant effects according to the subjective evaluation of patients - QIDS scale. c) response rate (50% reduction on the MADRS scale) and remission (MADRS ? 10). 2) time to return of depressive symptoms defined according to the criteria for the use of antidepressants within 12 weeks 3) safety profile of study medication Exploratory objectives: 1) Evaluate the antidepressant effect depending on: a) the intensity of acute psychological effects assessed using the subjective scale of 5D-ASCs and the objective scale of BPRS, b) depending on the retrospective assessment of persistent effects using the Persisting effects scale, c) the degree of eye contact with negative and neutral emotion faces measured by eye-tracking before and after treatment (on days 1 and 7). 2) To evaluate the neurobiology of the antidepressant effect in relation to: a) plasma levels of the major metabolite of psilocin, markers of neuroplasticity, antidepressant effect and stress (BDNF, prolactin, oxytocin, ACTH) at 90 min, 3, and 6 h after administration of study medication compared to pre-administration levels, b) changes in resting-state brain activity (connectivity, entropy) measured by simultaneous EEG / fMRI functional imaging methods before and after 1 and 7 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-65
2. Diagnosis of moderate to severe depressive disorder without psychotic symptoms - ICD-10 criteria F32.1-2 or F33.1-2 and at the same time MADRS score > 20
3. The duration of the current depressive episode is at least 3 months and maximum 2 years
4. Treatment-resistant depression defined as:

   1. Failure of at least 2 and at most 4 adequate treatments (6 weeks of full therapeutic dose of antidepressant or adequate non-pharmacological treatment - e.g. psychotherapy, neurostimulation treatment, phototherapy, etc.) within the current depressive episode, using at least 2 types of antidepressants with different pharmacological mechanisms of action (augmentation is taken as a second treatment) or
   2. Intolerance of 2 different treatments and 1 adequate treatment or
   3. Intolerance of 3 different antidepressant treatments.
5. Ability to understand the study protocol and to be able to complete all study visits and examinations as defined per protocol.
6. Participants in a clinical trial of childbearing potential must agree to the use of prescribed contraceptive methods for the duration of the study

Exclusion Criteria:

1. Severe psychiatric comorbidity (axis I MINI, ICD-10 F0.X - F99.X, the intensity of the disorder will be clinically assessed by the study clinician)
2. The current depressive phase is severe with psychotic symptoms (ICD-10: F32.3, F33.3)
3. MADRS suicidality score (item 10)> 4
4. Duration of the current depressive episode longer than 2 years
5. Current drug or alcohol dependence (ICD-10: F17.x) with the exception of tobacco and with the exception of abstinence lasting more than 2 years
6. Claustrophobia, inability to undergo MR examination
7. Pregnancy or breast-feeding or plan to become pregnant within the next 12 months
8. Intracranial hypertension, pulmonary hypertension, uncorrected arterial hypertension (BP> 150/100 mmHg)
9. Condition after stroke, myocardial infarction in the last 6 months
10. Heart failure
11. Untreated or decompensated hyperthyroidism
12. Glaucoma
13. Severe respiratory failure or acute respiratory depression
14. History of seizures
15. Other serious somatic disease or any other circumstance in which a significant increase in blood pressure would pose a serious threat to health (to be assessed by the study clinician)
16. Pacemaker
17. Metal implants made of MR incompatible materials
18. Regular use of medication that could interact with psilocybin (to be assessed by the investigator)
19. Regular use of antipsychotics with 5-HT2A receptor antagonist activity or discontinuation of their use for less than 14 days (eg risperidone, olanzapine, clozapine, quetiapine, ziprasidone)
20. Current use of monoamine oxidase inhibitors (MAOIs)
21. Previous experience with psilocybin, hallucinogenic mushrooms or ketamine is possible in a maximum of 10% of patients. This experience must not be during the last 12 months or during the current depressive episode.
22. Recent use of antidepressants with a direct antagonistic effect on 5-HT2A receptors such as SARI and tetracyclic antidepressants (eg trazodone, mirtazapine, mianserin) or discontinuation of their use for less than 14 days
23. Electroconvulsive therapy in the previous 3 months
24. Daily use of benzodiazepine anxiolytics higher than the equivalent of 10 mg diazepam
25. Allergy to any of the components of study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Verification of the rapid antidepressant effect of Psilocybin compared to Ketamine using the Montgomery-Asberg Depression Rating Scale at 24 hours post administration | 24 hours post drug administration
  The overall score of the Montgomery-Asberg Depression Rating Scale ranges from 0 to 60, a higher score indicates more severe depression.

SECONDARY OUTCOMES:
Comparing the response rate and duration of antidepressant effects of Psilocybin or Ketamine versus Midazolam (placebo) | At days 3, 7, 14, 21, 28, 35, 42, 56 and 84 post drug administration.
  Response rate defined as a 50% reduction on the Motgomery-Asberg Depression Rating Scale (range 0 to 60, a higher score indicates more severe depression).
Comparing the remission rate of depression after administration of Psilocybin or Ketamine versus placebo (Midazolam) | At days 3, 7, 14, 21, 28, 35, 42, 56 and 84 post drug administration.
  Remission (defined as a score of ≤10 on the Montgomery-Asberg Depression Rating Scale).
Comparing the time to return of depressive symptoms after administration of Psilocybin or Ketamine versus Midazolam (placebo) | At 12 weeks post drug administration.
  Return of depressive symptoms as defined by the clinical need to prescribe antidepressant medication by the study clinician. Criteria for the prescription of antidepressant medication are defined in the study protocol.
Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of 1 year.
  The safety of the study medications will be assessed by the analysis of the incidence of treatment-emergent adverse events
Comparing the response rate and duration of antidepressant effects of Psilocybin or Ketamine versus Midazolam (placebo) as rated by participants. | At days 1, 3, 7, 14, 21, 28, 35, 42, 56 and 84 post drug administration.
  Assessment via the Quick Inventory of Depressive Symptomatology (QIDS) which rates depression symptoms via self-assessment. Total QIDS scores range from 0 to 27 with higher scores indicating more severe depression.

OTHER OUTCOMES:
Assessment of the antidepressant effect in relation to the acute subjective psychological drug effects | At the end of dosing day, cca. 6 hours after drug administration
  Intesity of subjectively perceived acute psychological drug effects measured by the 5-Dimensional Altered States of Consciousness Rating Scale (5D-ASC)
Assessment of the antidepressant effect in relation to the acute objective psychological drug effects | At the end of dosing day, cca. 6 hours after drug administration
  Intesity of objectively perceived acute psychological drug effects measured by the Brief Psychiatric Rating Scale (BPRS). The BPRS consists of 18 items measuring the following factors: (1) anxiety, (2) emotional withdrawal, (3) conceptual disorganization, (4) guilt feelings, (5) tension, (6) mannerisms and posturing, (7) grandiosity, (8) depressive moods, (9) hostility, (10) suspiciousness, (11) hallucinatory behavior, (12) motor hyperactivity, (13) uncooperativeness, (14) unusual thought content, (15) blunted affect, (16) somatic concern, (17) excitement, and (18) disorientation. It uses a seven-item Likert scale with the following values: 1 = "not present", 2 = "very mild", 3 = "mild", 4 = "moderate", 5 = "moderately severe", 6 = "severe", 7 = "extremely severe".
Assessment of the antidepressant effect in relation to the retrospective assessment of persistent effects | At 1, 3, 6 and 12 months post drug administration.
  Persistent effects are measured by the Persistent Effects Questionnaire (A 143-item questionnaire detects information about changes in attitudes, moods, behavior, and spiritual experience that, on the basis of prior research (Pahnke 1969; Doblin 1991, Griffiths et al. 2006), is sensitive to the effects of psilocybin a month after the session.
Assessment of the antidepressant effect in relation to the degree of eye contact with negative and neutral emotional faces | Cca. 0.5 hours before and cca. 6 hours after treatment.
  Measured by eye-tracking.
Evaluate the neurobiology of the antidepressant effect in relation to plasmatic levels of Psilocin | 1.5 hours after drug administration
  Plasmatic levels of Psilocin, the major active metabolite of psilocybin will be measured in blood samples drawn from the participants.
Evaluate the neurobiology of the antidepressant effect in relation to plasmatic levels of Brain-Derived Neurotrophic Factor | Before drug administration (cca. 0.5 hours), then 1.5, 3 and 6 hours after drug administration.
  Changes of plasmatic concentrations of Brain-Derived Neurotrphic Factor (BDNF), a marker of neuroplasticity, will be measured in blood samples drawn from the participants.
Evaluate the neurobiology of the antidepressant effect in relation to plasmatic levels of Prolactine | Before drug administration (cca. 0.5 hours), then 1.5, 3 and 6 hours after drug administration.
  Changes of plasmatic concentrations of Prolactine, a marker of neuroplasticity, will be measured in blood samples drawn from the participants.
Evaluate the neurobiology of the antidepressant effect in relation to plasmatic levels of Oxytocine | Before drug administration (cca. 0.5 hours), then 1.5, 3 and 6 hours after drug administration.
  Changes of plasmatic concentration of Oxytocine, a marker of antidepressive effects, will be measured in blood samples drawn from the participants.
Evaluate the neurobiology of the antidepressant effect in relation to plasmatic levels of Adenocorticotropic Hormone. | Before drug administration (cca. 0.5 hours), then 1.5, 3 and 6 hours after drug administration.
  Changes of plasmatic concentration of Adenocorticotropic Hormone (ACTH), a marker of stress, will be measured in blood samples drawn from the participants.
Evaluate the neurobiology of the antidepressant effect in relation to plasmatic levels of Cortisol | Before drug administration (cca. 0.5 hours), then 1.5, 3 and 6 hours after drug administration.
  Changes of plasmatic concentration of Cortisol, a hormonal marker of stress, will be measured in blood samples drawn from the participants.
Evaluate the neurobiology of the antidepressant effect in relation to changes in resting state activity (connectivity, entropy) of the brain before and after drug administration. | Before (approx. 7 days) and after drug administration (1 and 7 days)
  Resting state activity will be evaluated by simultaneous fMRI + EEG.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health, Klecany, Czechia

IPD SHARING:
Plan to Share IPD: No